CLINICAL TRIAL: NCT01875640
Title: Decision Support for Parents Receiving Information About Child's Rare Disease
Acronym: DSD DST
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Virginia Commonwealth University (Other); Temple University (Other); University of California, Los Angeles (Other); Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, David E. Sandberg, PhD, Professor of Pediatrics, University of Michigan
Other Study IDs: 1360; 13-PAF00134 (Other: University of Michigan); HUM72007 (Other: University of Michigan)
Record Dates: First submitted 2013-05-30; First posted 2013-06-12 (Estimated); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Disorder of Sex Development; Intersex Conditions; Congenital Adrenal Hyperplasia; Hypospadias
Keywords: disorder of sex development; intersex; 46,XX congenital adrenal hyperplasia; hypospadias; decision support tool
MeSH Terms: conditions — Disorders of Sex Development; Adrenal Hyperplasia, Congenital; Hypospadias; Ovotesticular Disorders of Sex Development

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Usual Care: After obtaining consent, we will audio-record standard clinical consultations with specialists represented on the DSD team. These appointments will not utilize the Decision Support Tool. A qualitative analysis of these recordings will assess quality assurance and provide guidance for the development of the Decision Support Tool.
- Use of Decision Support Tool: After obtaining consent, we will audio-record standard clinical consultations with specialists represented on the DSD team. These appointments will utilize the Decision Support Tool (DST). A qualitative analysis of these recordings will assess the practicality of use and possible benefits of the DST's implementation.

SUMMARY:
The birth of a child with a disorder of sex development (DSD) is stressful for parents and members of the healthcare team. The "right" decisions about gender assignment (is it a boy? a girl?) and the best course of action (e.g., should there be surgery? what kind? when?) are not obvious. While there have been large advances in diagnostic assessments like genetic and endocrine testing, the tests do not always show what caused the DSD. And, even when the tests do reveal an explanation for the DSD, knowing what happened genetically or hormonally does not usually lead to a single "correct" treatment plan. Instead, it is likely that there are different acceptable treatment options - and parents will need to make decisions based, in part, on their personal preferences, values, and cultural background. Adding more stress to the situation is knowledge that many of the decisions that need to be made by parents early in a child's life are irreversible and exert life-long consequences for the child and the family.

To support parents becoming actively involved in making such decisions, and to reduce the likelihood of future worry and regret about decisions that have been made, the investigators will create a decision support tool (DST). The DST will help educate families about typical and atypical sex development of the body, the process by which DSD are diagnosed (especially how to interpret genetic test results), and possible relationships between diagnostic/genetic testing, decisions about care, and known consequences of those decisions on their child and entire family. The DST will be used by parents of young children together with their child's health care provider.

The investigators will bring together a network of researchers, health care providers, representatives of patient support and advocacy organizations, and parents of children with DSD to share their experiences. Participants of this network will be involved at each stage of creating the DST, revising it, and putting it into practice. At the end of this project, the investigators will have a fully formed DST that will be available for parents to use with their child's healthcare team as they are first learning their child may have a DSD.

ELIGIBILITY:
Inclusion Criteria:

* Must be a parent/caregiver of a patient who is newborn through 5 years old (i.e., 5.9 yrs).
* Patient clinical diagnosis of ambiguous genitalia (eg, 46,XX,Prader 2+; proximal hypospadias with uni/bilateral undescended testes) or sex chromosomes discordant with genital phenotype.
* Condition must be newly ascertained where decisions regarding surgical procedures (internal or external genitalia), diagnostic testing, and/or other aspects of clinical management have yet to be made.

Exclusion Criteria:

* Turner syndrome, Klinefelter syndrome, bladder or cloacal exstrophy.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: DSD
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2013-06; Primary Completion 2016-05 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
In-clinic communications | 2.5 years
  To assess characteristics of communications between parents/caregivers of young children with DSD and the children's healthcare providers by audio-recording standard-of-care appointments at DSD clinic.

CONTACTS AND LOCATIONS:
Overall Officials: David E Sandberg, PhD, Principal Investigator — University of Michigan
Locations (4):
- United States (4):
  - University of California Los Angeles, Los Angeles, California
  - University of Michigan, Ann Arbor, Michigan
  - Temple University, Philadelphia, Pennsylvania
  - Seattle Children's Hospital, Seattle, Washington